CLINICAL TRIAL: NCT00360867
Title: An Open Label Treatment Extension Study of AMG 706
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Amgen decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050130
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Solid Tumors
Keywords: Extension study; solid tumors
MeSH Terms: interventions — motesanib diphosphate

ARMS (1):
- 1 (Other): Single Arm
  Interventions: Drug: AMG 706

INTERVENTIONS:
Drug: AMG 706 — The dose of AMG 706 will be administered at the same dose level and schedule received at the conclusion of the previous study but will be no greater than 125 mg QD or 75 mg BID.
  Other Names: motesanib diphosphate

SUMMARY:
This is an extension study to provide ongoing treatment with AMG 706 monotherapy for subjects with solid tumors who have completed the planned duration of AMG 706 treatment on a separate Amgen protocol and have been evaluated as having stable disease or better. Subjects who are no longer eligible to continue AMG 706 treatment on a separate Amgen protocol (for reasons other than AMG 706 intolerance), but who are receiving clinical benefit or have the potential to receive clinical benefit from AMG 706 per the investigator are also eligible to participate in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 18 yrs or older with solid tumors, previously treated with AMG 706 on an Amgen protocol
* Subject must meet one of the following criteria: Subject has completed the planned duration of AMG 706 treatment on a separate Amgen protocol and has been evaluated as having stable disease or better or is no longer eligible to continue AMG 706 treatment on separate Amgen protocol for reasons other than AMG 706 intolerance, but is receiving clinical benefit from AMG 706 in the judgement of the investigator.
* Subject must meet one of the following criteria: Subject has received AMG 706 for at least 8 weeks or until the first protocol-specified tumor evaluation (whichever is longer) or
* Subject has received at least one dose of AMG 706 but did not receive AMG 706 for =/>8 weeks.
* Sign informed consent prior to study specific procedures.

Exclusion Criteria:

* Discontinued from prior AMG 706 study due to AMG 706-related adverse event including intolerance to AMG 706 or for any other reason that a subject's safety could be compromised with continued AMG 706 treatment.
* Has been off AMG 706 treatment >42 days prior to study day 1.
* Participating in any intervening investigational device or drug study between previous AMG 706 study and this AMG 706 study or is receiving any other investigational agent(s) other than AMG 706.
* Uncontrolled hypertension (resting blood pressure > 150/90 mmHg). Anti-hypertensive medications are allowed if the subject is stable on their current dose at time of study day1
* Requires additional systemic anticancer therapy for primary tumor.
* ANC < 1.0 x 10^9/L; PLT < 100 x 10^9/L; Hgb < 9 g/dL; serum creatinine > 2.0 mg/dL or calculated clearance < 40 mL/min; AST >2.5 x ULN, or AST =/> to or =/>5.0 x ULN if secondary to liver metastases; ALT >2.5 x ULN or ALT =/>5X ULN if liver metastasis are present; Alkaline phosphates >2.0 x ULN or =/>5 x ULN if liver and bone metastases are present; total bilirubin =/> 2 x ULN (except for subjects with UGT1A1 promoter polymorphism, ie, Gilbert's syndrome. Subjects enrolled with Gilbert's syndrome must have a total bilirubin <3 x ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2005-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety (serious adverse events, adverse events, blood pressure and laboratory tests) | Until objective evidence of disease progression, AMG 706 intolerance, or until loss of clinical benefit

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com